CLINICAL TRIAL: NCT05391178
Title: Improving Disease Severity in Alopecia Areata, Polymorphous Light Eruption, and Psoriasis Patients With Lumiton Technology
Brief Title: Improving Disease Severity
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00084854
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Psoriasis; Alopecia Areata; Polymorphous Light Eruption
MeSH Terms: conditions — Psoriasis; Alopecia Areata

STUDY DESIGN:
Intervention Model Description: A 12-week prospective pilot study involving a total of 15 patients, including five patients diagnosed with alopecia areata (AA), five patients diagnosed with polymorphous light eruption (PMLE), and five patients diagnosed with psoriasis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Psoriasis (Active Comparator): Psoriasis participants will be provided sleeves made from the Lumiton yarn to cover their arms. The participants will be instructed to wear the sleeves made from Lumiton yarn daily for 12 weeks both indoors and outdoors.
  Interventions: Other: Lumiton yarn sleeve
- Alopecia Areata (Active Comparator): Alopecia areata participants will be provided a hat made from the Lumiton yarn. The participants will be instructed to wear the hat made from Lumiton yarn daily for 12 weeks both indoors and outdoors.
  Interventions: Other: Lumiton yarn hat
- Polymorphous Light Eruption (Active Comparator): Polymorphous light eruption participants will be provided a shirt made from the Lumiton yarn. The participants will be instructed to wear the shirt made from Lumiton yarn daily for 12 weeks both indoors and outdoors.
  Interventions: Other: Lumiton yarn shirt

INTERVENTIONS:
Other: Lumiton yarn sleeve — Sleeve made from patented technology embedded in synthetic yarns that harnesses the sun's energy and generates red and near-infrared light - elevating apparel
  Arms: Psoriasis
Other: Lumiton yarn hat — Hat made from patented technology embedded in synthetic yarns that harnesses the sun's energy and generates red and near-infrared light - elevating apparel
  Arms: Alopecia Areata
Other: Lumiton yarn shirt — Shirt made from patented technology embedded in synthetic yarns that harnesses the sun's energy and generates red and near-infrared light - elevating apparel
  Arms: Polymorphous Light Eruption

SUMMARY:
Phototherapy, including ultraviolet B (UVB) and ultraviolet A (UVA) light, has been used to treat a number of dermatologic conditions. Psoriasis is one of the most common conditions treated with phototherapy, in which phototherapy is often indicated for extensive disease with contraindications for other systemic treatments. The mechanism of action of phototherapy for the treatment of psoriasis is not completely understood; however, it is known that UVB light induces apoptosis of pathogenic T cells and keratinocytes, which may reduce the overactive immune response and epidermal hyperproliferation. Phototherapy has shown some efficacy for other diseases, such as alopecia areata (AA) and polymorphous light eruption (PMLE). However, phototherapy is not always an accessible treatment option for patients due to cost or lack of time.

DETAILED DESCRIPTION:
Recent advancements in nanotechnology have led to the development of medical devices (lasers and LED devices) with unique phototherapy properties that emit radiation in the infrared wavelengths, allowing patients to benefit from the effects of phototherapy treatment in a more convenient way. Preclinical studies demonstrated the positive effects of infrared radiation exposure on the skin including, increased collagen synthesis and expression of transforming growth factor-beta1 (TGF-beta1). Other studies suggested possible antimicrobial effects from infrared radiation, with decreased colonization of Staphylococcus aureus, Escherichia coli, and Klebsiella pneumoniae on the skin after exposure. Compared to other fabric technology, such as Far-Infrared (FIR) fabric technology that reflects body heat, fabric made from Lumiton yarn converts external light in the UV and visible spectrum and emits light in the red and near-infrared spectrum for the body. Lumiton yarn absorbs energy from 350 nm to 600 nm (the light spectrum from UV to visible red light) and emit energy from 600 to 1000 nm (red, near-infrared spectrum). The Lumiton yarn contains red/NIR light-emitting dyes. The effectiveness of the technology is proportional to the intensity of the light, with its peak effectiveness under sunlight.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants ≥18 years of age
* Participants who live in the US,
* Participants who are diagnosed with mild-to-severe AA, PMLE, or psoriasis
* Participants have sufficient command of the English language

Exclusion Criteria:

* Participants less than the age of 18
* Participants who do not live in the US
* Participants who are not diagnosed with mild to severe AA, PMLE, or psoriasis
* Participants without a sufficient command of the English language
* Participants with concurrent medical conditions that are at risk of confounding the study outcomes
* Participants currently using concomitant phototherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Disease severity - photo | Baseline
  Lesion photos
Disease severity - photo | Week 12
  Lesion photos
Disease severity - PASI | Baseline
  Psoriasis Area and Severity Index-75 (PASI-75%) scores The percentage area affected by psoriasis is evaluated in the four regions of the body. In each region, the area is expressed as nil (0), 1-9% (score 1), 10-29% (score 2), 30-49% (score 3), 50-69% (score 4), 70-89% (score 5) or 90-100% (score 6).
Disease severity - PASI | Week 12
  Psoriasis Area and Severity Index-75 (PASI-75%) scores The percentage area affected by psoriasis is evaluated in the four regions of the body. In each region, the area is expressed as nil (0), 1-9% (score 1), 10-29% (score 2), 30-49% (score 3), 50-69% (score 4), 70-89% (score 5) or 90-100% (score 6).
Disease severity - SALT | Baseline
  Severity of Alopecia Tool (SALT) score The SALT score is computed by measuring the percentage of hair loss in each of 4 areas of the scalp-vertex (40%), right profile (18%), left profile (18%), and posterior (24%)-and adding the total to achieve a composite score.
Disease severity - SALT | Week 12
  Severity of Alopecia Tool (SALT) score The SALT score is computed by measuring the percentage of hair loss in each of 4 areas of the scalp-vertex (40%), right profile (18%), left profile (18%), and posterior (24%)-and adding the total to achieve a composite score.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Jorizzo, M.D., Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Dermatology, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
This is pilot research, there is no decision to share individual participant data

REFERENCES:
- [Background] Barros NM, Sbroglio LL, Buffara MO, Baka JLCES, Pessoa AS, Azulay-Abulafia L. Phototherapy. An Bras Dermatol. 2021 Jul-Aug;96(4):397-407. doi: 10.1016/j.abd.2021.03.001. Epub 2021 Apr 2. PMID 33849754
- [Background] Tsai SR, Hamblin MR. Biological effects and medical applications of infrared radiation. J Photochem Photobiol B. 2017 May;170:197-207. doi: 10.1016/j.jphotobiol.2017.04.014. Epub 2017 Apr 13. PMID 28441605
- [Background] Toyokawa H, Matsui Y, Uhara J, Tsuchiya H, Teshima S, Nakanishi H, Kwon AH, Azuma Y, Nagaoka T, Ogawa T, Kamiyama Y. Promotive effects of far-infrared ray on full-thickness skin wound healing in rats. Exp Biol Med (Maywood). 2003 Jun;228(6):724-9. doi: 10.1177/153537020322800612. PMID 12773705
- [Background] Chung J, Lee S. Development of nanofibrous membranes with far-infrared radiation and their antimicrobial properties. Fibers and Polymers. 2014;15(6).